CLINICAL TRIAL: NCT02249949
Title: A Phase II Study of the Peroxisome Proliferator-Activated Receptor Gamma Agonist, Efatutazone in Patients With Previously Treated, Unresectable Myxoid Liposarcoma
Brief Title: Efatutazone Dihydrochloride in Treating Patients With Previously Treated Myxoid Liposarcoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A091202; NCI-2014-01028 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Liposarcoma
MeSH Terms: conditions — Liposarcoma | interventions — efatutazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- efatutazone dihydrochloride (Experimental): Patients receive efatutazone dihydrochloride PO BID continuously. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: efatutazone

INTERVENTIONS:
Drug: efatutazone — Given PO

SUMMARY:
This phase II trial studies how well efatutazone dihydrochloride works in treating patients with previously treated myxoid liposarcoma that cannot be removed by surgery. Drugs used in chemotherapy, such as efatutazone dihydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the confirmed response rate for efatutazone dihydrochloride (efatutazone) in patients with advanced myxoid liposarcoma whose disease has progressed on at least one prior therapy.

SECONDARY OBJECTIVES:

I. To assess the progression free survival (PFS), overall survival (OS), and adverse event rates for efatutazone treated patients with advanced myxoid liposarcoma whose disease has progressed on at least one prior therapy.

TERTIARY OBJECTIVES:

I. To assess the predictive value of peroxisome proliferator-activated receptor (PPAR) and retinoid X receptors (RXR) tumor expression from archived patient tumor samples.

II. To assess the predictive value of the expression of PPARgamma-regulated markers of adipocytes differentiation.

III. To assess the predictive value of the expression of PPARgamma-regulated cell cycle proteins.

IV. To assess the effects of efatutazone treatment on serum adiponectin levels.

OUTLINE:

Patients receive efatutazone dihydrochloride orally (PO) twice daily (BID) continuously. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 2 years and then every 6 months for up to 5 years.

ELIGIBILITY:
* Patients must have a formalin-fixed, paraffin-embedded (FFPE) tumor block OR 1 representative hematoxylin and eosin (H&E) and 20 unstained myxoid liposarcoma tissue slides available for submission to central pathology review; this review is mandatory prior to registration to confirm eligibility
* Measurable disease
* Progression on at least one prior systemic chemotherapy for advanced, unresectable or metastatic disease; prior adjuvant or neoadjuvant therapy is not included as prior systemic chemotherapy unless treatment occurred within the 6 months prior to study enrollment

  * There is no limit to the number of prior lines of treatment a patient has received
  * No treatment with biologic therapy, immunotherapy, chemotherapy, investigational agent for malignancy, or radiation =< 28 days before study registration; no treatment with nitrosourea or mitomycin =< 42 days before study registration
  * Patients should have resolution of any toxic effects of prior therapy (except alopecia) to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0, grade 1 or less
* No history of the following:

  * Class III or IV congestive heart failure (CHF)
  * Pericardial effusion =< 12 months (grade 3 or 4)
  * Pericardial involvement with tumor
  * Grade 2 or higher pleural effusion =< 6 months
* No symptomatic, untreated, or uncontrolled brain metastases present
* Not pregnant and not nursing; for women of childbearing potential only, a negative pregnancy test done =< 7 days prior to registration is required; a female of childbearing potential is a sexually mature female who:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Patients with diabetes mellitus requiring concurrent treatment with insulin or thiazolidinedione (TZD) oral agents are not eligible
* Patients with known hypersensitivity to any TZD oral agents are not eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelet count >= 75,000/mm^3
* Creatinine =< 1.5 mg/dL x upper limits of normal (ULN) OR calculated (calc.) creatinine clearance >= 30 mL/min
* Bilirubin =< 1.5 x ULN; for subjects with liver metastases =< 3 x ULN is allowed
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN; for subjects with liver metastases, SGOT (AST) and SGPT (ALT) < 5 x the upper normal limit of institution's normal range is allowed
* Eligible patients must have histopathologically confirmed myxoid liposarcoma with confirmation of DDIT3 rearrangement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pishvaian, MD, PhD, Study Chair — Georgetown University
Locations (127):
- United States (127):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Memorial and Saint Elizabeth's Health Care Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Integris Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A protocol amendment (Update #02) removed the option for patients to be randomized to Placebo; the study went from being a randomized study to a single arm study. The discrepancy in the number of patients who 'Started' the study and the Protocol Enrollment number is due to there being 2 patients randomized to Placebo prior to Update #02.
Period: Overall Study
Arm/Group | Efatutazone Dihydrochloride
Started | 13
Completed | 11
Not Completed | 2
Not completed — Cancelled prior to treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Efatutazone Dihydrochloride
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 6
    1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate Per the RECIST 1.1 Criteria
Description: The response rate (percentage) is the percent of patients whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients.
Time Frame: Up to 24 weeks (8 cycles)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Efatutazone Dihydrochloride
Number analyzed (Participants) | 11
percentage of patients | 0 [0 to 28]

2. Secondary Outcome: Progression Free Survival (PFS) Determined Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Description: Progression free survival (PFS) is defined as the time from study entry to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from study entry to the first of either disease progression or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efatutazone Dihydrochloride
Number analyzed (Participants) | 11
months | 1.4 [1.2 to NA] — The 95% confidence interval upper limit was not obtained.

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from study entry to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from study entry to death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Efatutazone Dihydrochloride
Number analyzed (Participants) | 11
months | 8.6 [6.8 to NA] — The 95% confidence interval upper limit was not obtained.

4. Secondary Outcome: Incidence of Grade 3+ Adverse Events Summarized Using Common Terminology Criteria for Adverse Events Version 4.0
Description: Incidence of grade 3+ adverse events summarized using Common Terminology Criteria for Adverse Events version 4.0: The frequency and percentage of grade 3+ adverse events will be estimated
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Efatutazone Dihydrochloride
Number analyzed (Participants) | 11
Participants
  at least one grade 3 or worse AE | 6
  at least one grade 4 or worse AE | 3

ADVERSE EVENTS:
Time Frame: Adverse events are assessed weekly during cycle 1, and then on day 1 (+/- 4 days) for cycles 2-4; then day 1 (+/- 7 days) of every odd numbered cycle for Cycle 5 and beyond; up to 5 years.
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for completed patients. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Efatutazone Dihydrochloride
All-Cause Mortality (participants affected / at risk) | 8/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efatutazone Dihydrochloride (N=11)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Edema trunk (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efatutazone Dihydrochloride (N=11)
Anemia (Blood and lymphatic system disorders) | 6 (19)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (2)
Edema limbs (General disorders) | 8 (26)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (21)
Cholesterol high (Investigations) | 1 (2)
Creatinine increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (5)
Neutrophil count decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 8 (23)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (4)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (4)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT02249949/Prot_SAP_000.pdf